CLINICAL TRIAL: NCT04147676
Title: Multicentre Trial to Assess the Performance of Centralized Assay Solutions for Detection of MTB and Resistance to Rifampin and Isoniazid
Brief Title: Evaluation of Centralised TB Assay Solutions
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 7213-2/1
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2019-10

CONDITIONS: Tuberculosis; Drug-resistant Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum specimens M. tuberculosis cultures isolates from patient specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TB suspects: Sputum specimens will be collected from TB suspects enrolled in the study.
  The specimens will be tested with
  1. Roche cobas MTB - for the detection of Mycobacterium tuberculosis complex
  2. Roche cobas MTB-RIF/INH - all specimens that are Mycobacterium tuberculosis complex positive will be reflexed to the Roche cobas MTB-RIF/INH test for the detection of resistance to rifampicin and isoniazid
  3. Hain FluoroType MTBDR - for the detection of Mycobacterium tuberculosis complex and the detection of resistance to rifampicin and isoniazid

SUMMARY:
Tuberculosis (TB) remains a life-threatening disease partly due to increasing incidence of multidrug and extensively drug-resistant TB. Diagnostic based on culture and conventional drug susceptibility testing using media take several weeks leading to prolonged periods of ineffective therapy and ongoing transmission. Development of rapid molecular diagnostic tests for the identification of Mycobacterium tuberculosis (MTB) and drug resistance has become a high priority.

The Xpert® MTB/RIF Assay does not provide information on INH-resistance and the LPA is only recommended for use in smear-positive samples, complex to perform and requires manual interpretation. Several novel assays have been recently developed/CE-marked offering high sample throughput and higher sensitivity for detection of MTB, RIF- and INH-resistance in centralized laboratories. However, published data on their performance and operational characteristics is extremely limited.

This is a prospective, multicentre, diagnostic accuracy trial in which the performance of centralised TB assay solutions will be assessed at the intended setting of use with culture, phenotypic DST and sequencing as reference standard.

Potential trial participants will be identified at participating TB clinics or hospitals (enrolment sites). Sputum samples will be collected and transported to the associated TB reference laboratories (testing sites).

In order for the results of this trial to be generalizable, adults with symptoms compatible with pulmonary TB undergoing evaluation will be screened for inclusion at geographically diverse participating centres in high burden TB countries. Additionally, to supplement the drug-resistant cases to timely achieve accurate performance estimates, well-characterized frozen sputum samples from the FIND specimen bank will be used.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included as trial participants only if all of the following inclusion criteria apply:

* Aged ≥18 years
* Clinical suspicion of pulmonary TB including cough ≥2 weeks (or any duration if HIV positive ) and ≥1 other symptom typical of pulmonary TB listed below:

  * Fever
  * Malaise
  * Recent weight loss
  * Night sweats
  * Contact with active case
  * Haemoptysis
  * Chest pain
  * Loss of appetite

Exclusion Criteria:

Participants are excluded from the trial if any of the following exclusion criteria apply:

* Unwilling or unable to provide informed consent
* Unwilling to provide four sputum specimens at enrolment i.e. 2x sputa on day 1 and 2x sputa on day 2 (up to 1 week from enrolment)
* Patients with only extra-pulmonary TB signs & symptoms
* Receipt of any dose of TB treatment within 6 months prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom pulmonary TB is suspected. Additionally, well-characterized RIF-resistant and INH-resistant samples will be used to supplement drug-resistant cases.
Sampling Method: Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy for MTB detection | four to six months
  clinical sensitivity and specificity by smear-status measured against mycobacterial culture as the reference standard.
Diagnostic accuracy for RIF/INH detection | four to six months
  clinical point estimates of sensitivity and specificity measured against a composite reference standard of phenotypic DST and targeted sequencing.

SECONDARY OUTCOMES:
Operational characteristics: | four to six months
  description of operator experience with the assays through daily observed usage and user appraisal questionnaires.

CONTACTS AND LOCATIONS:
Locations (6):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- Forschungszentrum Borstel. Leibniz Lungenzentrum (Borstel), Borstel, Germany
- India (2):
  - Indian Council of Medical Research (ICMR) Regional Medical Research Centre, Bhubaneswar
  - National Institute for Research in Tuberculosis, Chennai
- Institute of Phthisiopneumology "Ch. Draganiuc" (PPI NRL), Moldova, Chisinau, Moldova
- Division of Wits Health Consortium (DMMH), Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Undecided